

# TRANSLATIONAL STATISTICAL ANALYSIS PLAN KTE-C19-108 TRANSLATIONAL ANALYSIS

| Sponsor: | Kite Pharma, Inc. 2400 Broadway Santa Monica, CA 90404 United States of America |
|---|---|
| <b>Product Name:</b> | KTE-X19 |
| Protocol Title: | A Phase 1 Multicenter Study Evaluating the Safety and Tolerability of KTE-X19 in Adult Subjects with Relapsed/Refractory Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma |
| <b>Protocol Number</b> | KTE-C19-108 (ZUMA-8) |
| Version Number: | Version 1.05 |
| Release Date: | 24 September 2021 |
| Replaces Previous<br>Version(s): | |

#### **CONFIDENTIALITY NOTICE**

This document contains confidential information of Kite Pharma Inc., a wholly owned subsidiary of Gilead Sciences Inc. This document must not be disclosed to anyone other than the site research staff, collaborators, and members of the Institutional Review Board/Independent Ethics Committee, a scientific review board or an equivalent. The information in this document cannot be used for any purpose other than the conduct of the clinical investigation without the prior written consent of Kite Pharma Inc. Questions regarding how this document should be used or the conduct of the clinical trial should be directed to the key sponsor contacts.

## **TABLE OF CONTENTS**

| TA | BLE O | F CONTE | NTS | 2 |
|---|---|---|---|---|
| LIS | T OF T | ABLES | | 2 |
| LIS | T OF A | BBREVL | ATIONS | 3 |
| 1. | | | ON | |
| 2. | | | | |
| 2. | 2.1. | | ves | |
| | 2.1. | | esis | |
| 3. | ENDI | POINTS, S | SUBGROUPS AND COVARIATES | 6 |
| | 3.1. | Dataset | s to be Included | 6 |
| | 3.2. | Endpoir | nts | 7 |
| | 3.3. | Outcom | nes, Subgroups, and Covariates | 7 |
| 4. | DEFI | NITIONS | | 8 |
| | 4.1. | | | |
| | 4.2.<br>4.3. | • | | |
| | 4.4. | | easurements of Product Characteristics. | |
| 5. | ANA | LYSIS SE | TS | 10 |
| | | | ANALYSIS | 11 |
| | 6.1. General Methods | | | 11 |
| | 6.2. | | s | |
| | | 6.2.1. | Characterize the anti-CD19 CAR T Cell Expansion (PK) and Serum | 11 |
| | | 6.2.2. | Cytokine Profile | |
| | | 6.2.3. | Explore MRD negativity | |
| 7. | APPE | ENDIX | | 12 |
| | 7.1. | Definiti | on of Analytic Visit Windows for CAR T Cells in Blood | 12 |
| | 7.2. | Definiti | on of Analytic Visit Windows for Cytokines in Serum | 12 |
| | 7.3. | Using T | rapezoidal Rule to Approximate the Area under the Curve (AUC) | 13 |
| | | | LIST OF TABLES | |
| | Table | 3-1. | Data Overview on Assay Methods and Biomarker Lists | 6 |
| | Table | - | Analytic Visit Windows for CAR T Cells in Blood | 12 |
| | Table | 7-2. | Analytic Visit Windows for Cytokines in Serum | 12 |

#### LIST OF ABBREVIATIONS

AUC Area under the curve
CAR Chimeric antigen receptor
CD Cluster of differentiation
CRP C-reactive protein

CRS Cytokine release syndrome
CXCL C-X-C motif chemokine ligand

ddPCR Droplet digital polymerase chain reaction

DLT Dose-limiting toxicity
DNA Deoxyribonucleic acid

ICAM Intercellular adhesion molecule

IFN Interferon IL Interleukin

LOQ Limit of quantification
LYMLE Lymphocyte (%)
MONOLE Monocyte (%)

MRD Minimal residual disease MTD Maximum toxicity dose

PBMC Peripheral blood mononuclear cells

PD Pharmacodynamics PK Pharmacokinetic

SAP Statistical analysis plan
TNF Tumor necrosis factor

TSAP Translational statistical analysis plan VCAM Vascular cell adhesion molecule

WBC White blood cell count

#### 1. INTRODUCTION

This translational statistical analysis plan (TSAP) outlines the analyses to be conducted for pharmacokinetics (PK) (levels of anti-CD19 CAR T cells), pharmacodynamics (levels of cytokines and other key analytes) and product characteristics data for Study KTE-C19-108 (ZUMA-8) titled "A Phase 1 Multicenter Study Evaluating the Safety and Tolerability of KTE-X19 in Adult Subjects with Relapsed/Refractory Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma", as described in protocol amendment 3 dated 01 September 2021.

## 2. OBJECTIVES

## 2.1. Objectives

- Characterize the anti-CD19 CAR T cell expansion (PK)
- Characterize profile for selected serum cytokines (PD)
- Characterize the product characteristics
- Characterize Minimal Residual Disease (MRD) data for bone marrow and peripheral blood samples

## 2.2. Hypothesis

The analyses outlined in this TSAP are CCI and and no formal pre-specified hypothesis will be tested.

# 3. ENDPOINTS, SUBGROUPS AND COVARIATES

#### 3.1. Datasets to be Included

Table 3-1. Data Overview on Assay Methods and Biomarker Lists

| Data type | Assay Method/<br>Sample type | Biomarker Set | Assessment Time<br>Points |
|---|---|---|---|
| CCI | | | |
| | | | CCI |
| Product<br>characteristics | | Total T Cells (106), CD3 Cells (total number and %), CD4 Cells (total number and % of viable CD3+ cells), CD8 Cells (total number and % of viable CD3+ cells), CD4/CD8 Ratio, Central Memory Cells (total number and % of viable CD3+ cells), Effector Cells (total number and % of viable CD3+ cells), Effector Memory Cells (total number and % of viable CD3+ cells), Interferon Gamma level (pg/mL), Naïve Cells (total number and % of viable CD3+ cells), Total CAR+ T cells (106), Transduction Rate (%), Viability (%), Vector Copy Number, CCR7+ (Tnaive + Tcm) % and number, CCR7- (Tem + Teff) % and number. | |
| CCI | | | |

## 3.2. Endpoints

- Levels of anti-CD19 CAR T cells in blood samples measured as anti-CD19 CAR+ cells/μL by visit, peak, area under the curve (AUC) (from infusion to Day 28), and time-to-peak (details for the derivations are included in the definition Section 4.2)
- Levels of cytokines in serum by visit, change from baseline at Day 0, Day 1, Day 4 and Day 7, fold change from baseline at Day 0, Day 1, Day 4 and Day 7, peak, Day 0 Day 28 AUC, and time to peak (details for the derivations are included in the definition Section 4.3)
- Product attributes measurements after product manufacturing and prior to dosing
- Levels of CLL of nucleated cells and of CD45+Lymphocytes by visit, Screening, Bridging Chemotherapy, Day 28, Month 3

## 3.3. Outcomes, Subgroups, and Covariates

No outcomes, subgroups and covariates will be used for analyses in this TSAP.

#### 4. **DEFINITIONS**

#### 4.1. General

**Study Day 0:** defined as the day the subject received the first KTE-X19 infusion.

**Baseline:** the baseline value is defined as the last value taken prior to first dose of conditioning chemotherapy. If the enrolled subjects do not receive conditioning chemotherapy, the baseline value is defined as the last value taken prior to enrollment/leukapheresis.

## 4.2. Key Measurements of Anti-CD19 CAR+ T Cell

The presence, expansion, and persistence of anti-CD19 CAR T cells in peripheral blood will be measured by ddPCR analysis.

**Scheduled blood draw for anti-CD19 CAR T cell:** This TSAP will focus on the anti-CD19 CAR T cell data collected as per planned assessment, based on the analysis visits defined in Appendix Section 7.1.

Baseline number of anti-CD19 CAR T cells (cells/ $\mu$ L) is defined as 0 before the KTE-X19 infusion on Day 0, and number of CAR T (cell/ $\mu$ L) will not be derived.

#### Number of anti-CD19 CAR T (cells/ µL) derivation:

#### **Derivation 1**

- Alpha =  $(CAR / \mu g DNA \text{ at timepoint}) / 162,000$
- Beta =  $(CAR / \mu g DNA \text{ of product } / 162,000) / \%$  Transduction (by flow of product)
- Optimized % CAR+ PBMC = (Alpha/Beta)
- Number of anti-CD19 CAR T (cells/µL blood) is defined as:

1000\*(WBC [10^9/L])\*(MONOLE [%] + LYMLE [%])/100\*Optimized %CAR+PBMC

**Peak of anti-CD19 CAR T cell (cells/ μL blood)** is defined as the maximum absolute number of anti-CD19 CAR T (cells/ μL) in serum attained after Day 0.

**Time to Peak of anti-CD19 CAR T cell** is defined as the number of days from Day 0 to the day when the peak of anti-CD 19 CAR T cell was attained as "Peak date – KTE-X19 Dosing date + 1."

Area-Under-Curve (AUC) of level of anti-CD19 CAR T cell (cells/μL • days) from Day 0 to Day 28 is defined as the AUC in a plot of levels of anti-CD19 CAR T cells against scheduled visits from Day 0 to Day 28. This AUC measures the total levels of anti-CD19 CAR T cells over time. Given the anti-CD19 CAR T cells are measured at certain discrete time points, the trapezoidal rule will be used to estimate the AUCs.



#### 4.4. Key Measurements of Product Characteristics

All product characteristics as defined in Table 3-1 will be summarized individually.

In addition to all the measured product characteristics, the following additional analytes will be derived:

• 2 additional analytes will be derived for exploration:

CD4/CD8 Ratio is defined as: 
$$\frac{\text{CD4 Cells (\%)}}{\text{CD8 Cells (\%)}}$$

IFN-gamma/Transduction rate is defined as: Interferon-gamma normalized by transduction rate

Interferon gamma level in product
Transduction rate

## 5. ANALYSIS SETS

Translational analysis will use the analysis sets defined in clinical SAP unless otherwise specified. The following subjects will be involved in analysis:

## Safety Analysis Set

The safety analysis set is defined as all subjects treated with any dose of KTE-X19. The safety analysis set will be the primary analysis set used to summarize the translational data in this TSAP.

## 6. STATISTICAL ANALYSIS

#### 6.1. General Methods

The following methods will be applied to the data analysis when applicable.

#### Summary statistics

Summary statistics refers to the number of subjects, median, 1<sup>st</sup> quartile (Q1), 3<sup>rd</sup> quartile (Q3), minimum, and maximum for continuous measurements in overall and by cohorts.



#### **6.2.2.** Characterize Product Attributes

- The safety analysis set will be used to summarize the product characteristics data.
- Summary statistics will be generated in overall data and by cohorts.



# 7. APPENDIX



# 7.3. Using Trapezoidal Rule to Approximate the Area under the Curve (AUC)



AUC 
$$\approx \frac{1}{2}(y_0 + y_1) \cdot \Delta x + \frac{1}{2}(y_1 + y_2) \cdot \Delta x + \frac{1}{2}(y_2 + y_3) \cdot \Delta x + \dots$$